CLINICAL TRIAL: NCT05052879
Title: National, Multicenter, Randomized, Double-blind, Double-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Toronto Association in the Treatment of Erectile Dysfunction and Premature Ejaculation
Brief Title: Efficacy and Safety of Toronto Association in the Treatment of Erectile Dysfunction and Premature Ejaculation
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0220 - TORONTO
Record Dates: First submitted 2021-09-14; First posted 2021-09-22 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Erectile Dysfunction; Premature Ejaculation
Keywords: Erectile dysfunction; Premature Ejaculation
MeSH Terms: conditions — Erectile Dysfunction; Premature Ejaculation | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TORONTO 20 + 30/60 (Experimental): The study is double-dummy. The patient must take 2 tablets before the sexual intercourse, as follows:
  1 tablet of Toronto association, oral;
  1 tablet of tadalafil placebo, oral.
  Interventions: Drug: Toronto association; Other: Tadalafil placebo
- TADALAFIL (Active Comparator): The study is double-dummy. The patient must take 2 tablets before the sexual intercourse, as follows:
  1 tablet of tadalafil , oral;
  1 tablet of Toronto association placebo, oral.
  Interventions: Drug: Tadalafil; Other: Toronto association placebo

INTERVENTIONS:
Drug: Toronto association — Toronto association coated tablet, 20 mg + 30 mg or 20 mg + 60 mg, oral, 2 hours before the sexual intercourse.
  Arms: TORONTO 20 + 30/60
Drug: Tadalafil — Tadalafil coated tablet, 20 mg, oral, 2 hours before the sexual intercourse.
  Arms: TADALAFIL
Other: Tadalafil placebo — Tadalafil placebo coated tablet, oral, 2 hours before the sexual intercourse.
  Arms: TORONTO 20 + 30/60
Other: Toronto association placebo — Toronto association placebo coated tablet, oral, 2 hours before the sexual intercourse.
  Arms: TADALAFIL

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Toronto association in the treatment of both sexual dysfunction: erectile dysfunction and premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Male participants, with age greater than or equal to 18 years;
* Heterosexual, sexually active participants in a stable and monogamous relationship for at least 6 months before screening and who plan to maintain this relationship throughout the study period;
* Participants with erectile dysfunction, in stable and effective treatment with PDE-5 inhibitors;
* Participants diagnosed with premature ejaculation;
* Participants with IELT ≤ 2 minutes;
* Participants with score ≥ 25 points in the erectile function questionnaire;
* Participants (or partners) who use at least one contraceptive method.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participation in a clinical trial in the year prior to this study;
* Known hypersensitivity to any of the formula compounds;
* Participants with cardiovascular disease for whom sexual activity is inadvisable
* History or current experience of surgical interventions or radiotherapy in the pelvic region, neurological conditions, trauma or infections that are associated with the symptoms premature ejaculation;
* Diagnosis of other diseases or conditions in the urinary tract;
* Participants with conditions that may predispose them to priapism;
* History of severe psychiatric or psychosocial disorders;
* Participant whose partner has clinically important sexual dysfunctions.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment response after 4 weeks of treatment. | 4 weeks
  The treatment response will be based on the participant's questionnaire answer after the treatment.
Percentage of participants with treatment response after 8 weeks of treatment. | 8 weeks
  The treatment response will be based on the participant's questionnaire answer after the treatment.

SECONDARY OUTCOMES:
Adverse events | 103 days
  Incidence and severity of adverse events recorded during the study.

IPD SHARING:
Plan to Share IPD: No